CLINICAL TRIAL: NCT04064632
Title: Multicenter, National, Prospective, Open Label, Randomized, Pilot, Proof-of-concept Study on the Use of Rilpivirine Plus Darunavir/Cobicistat as Substitutive Agents in Virologic Suppressed Patients
Brief Title: RPV+DRV/Cobi Dual Therapy in Subjects With HIV Controlled Infection
Acronym: PROBE2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: San Raffaele University Hospital, Italy (Other)
Responsible Party: Principal Investigator, Franco Maggiolo, Managing Director, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG23-1
Record Dates: First submitted 2019-08-13; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: HIV Infection
Keywords: Switch therapy; HIV; Dual ART; Rilpivirine; Darunavir/cobicistat; NNRTI; PI; virologically suppressed patients
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine; Darunavir; Cobicistat

STUDY DESIGN:
Intervention Model Description: Patients are randomly allocated into two arms:
  The control arm continues the baseline therapy based on 3 drugs (2 NRTIs) for 24 weeks and then will be switched to receive rilpivirine and cobicistat/darunavir co-formulated tablets (a tablet day).
  The experimental arm receives rilpivirine and cobicistat/darunavir coformulated tablets at randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPV +DRV/cobi (Experimental): The experimental receives rilpivirine (a tablet/day) and cobicistat/darunavir co-formulated tablets (a tablet day) since randomization.
  Interventions: Drug: Rilpivirine + darunavir/cobicistat
- baseline therapy (CAR) (Active Comparator): The control arm continues the baseline therapy (CAR) based on 3 drugs (2 NRTIs) for 24 weeks and then will be switched to receive rilpivirine (a tablet/day) and cobicistat/darunavir co-formulated tablets (a tablet day).
  Interventions: Drug: Rilpivirine + darunavir/cobicistat

INTERVENTIONS:
Drug: Rilpivirine + darunavir/cobicistat — Switch to a dual ART

SUMMARY:
This study evaluates efficacy and safety of rilpivirine as substitutive agent for the nucleosidic backbone of HAART in virologic suppressed patients when combined with cobicistat-boosted darunavir.

DETAILED DESCRIPTION:
HAART is generally based on the combination of three active drugs. Two of them, usually defined the backbone, belong to the nucleosidic analogues class (NRTI). In the last years, drugs of this class have been associated to several long-term adverse events of HAART such as lipoatrophy, cardiovascular diseases, bone and kidney toxicity. Furthermore the need of a triple drug regimen has recently been questioned as maintenance therapy in well controlled chronically treated subjects. In this setting, less drug regimens (LDR) have been proposed. LDR would allow a reduced exposure to drugs and eventually limit drug-drug interactions, drug-related toxicities and would allow treatment simplification so to enhance HAART acceptability, tolerability and persistence.

ELIGIBILITY:
Inclusion Criteria:

1. Written signed and dated informed consent to participate in the study must be given by the subject, in accordance with the International Conference of Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E627 and applicable regulations, before completing any procedure related to the study.
2. HIV-1 documented infection
3. Male and female subjects > 18 years of age.
4. Males, or non-pregnant, non-lactating females of childbearing potential, as demonstrated by a negative pregnancy test, who agree to comply with any applicable contraceptive requirements of the protocol. Women of child-bearing potential with a negative pregnancy test at Screening and Day 1 should agree to use one of the following methods: Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IMP, throughout the study, and for at least 2 weeks after; Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide) IUD and male condom Male partner sterilization confirmed and male condom Approved hormonal contraception and male condom Any other method with published data showing that the expected failure rate is <1% per year and use male condo Any contraception method must be used for at least 2 weeks after discontinuation of IMP.
5. Being on a stable therapy for at least 6 months.
6. SBR must be based on any 2NRTI plus a third NNRTI, PI or INI agent. Any possible registered drug is allowed among NRTI (e.g. tenofovir, lamivudine, emtricitabine and abacavir), PI (e.g. lopinavir, atazanavir, darunavir), NNRTI (efavirenz, nevirapine, rilpivirine) or INI (raltegravir, elvitegravir, dolutegravir).
7. Having a fully suppressed HIV replication as documented by 2 prior HIV-RNA tests (at least two months apart) below the detection limit (50 copies/ml).
8. Subjects and investigator must agree that participation in this study is in the best interest of the subject.

Exclusion Criteria:

1. Patients co-infected with HBV
2. Pregnancy or breast feeding.
3. Positive anamnesis for allergy to NNRTI
4. A positive historical genotypic test showing resistance-inducing mutation either toward NNRTIs or PIs
5. History or other evidence of severe illness (malignancy or OI) requiring active treatment and/or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
6. Anticipated need for Hepatitis C virus (HCV) therapy during the study period
7. Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses
8. All conditions and medicinal products listed in contraindications of DRV/c and rilpivirine
9. Subjects with current or prior (previous year) history of alcohol or other substance abuse.
10. Patients who have previously been screened for or enrolled into this study and subsequently withdrawn.
11. Patients having been given investigational drugs within 12 weeks prior to screening.
12. Inability or unwillingness to provide informed consent.
13. Life expectancy < 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
clinical response | 24 weeks
  proportion of patients with HIV-RNA < 50 copies/ml (FDA snapshot)
Virological response | 24 weeks
  proportion of patients with HIV-RNA > 50 copies/ml (FDA snapshot)
clinical response | 48 weeks
  proportion of patients with HIV-RNA < 50 copies/ml

SECONDARY OUTCOMES:
Tolerability (number and proportion of AEs) | 24 weeks
  AEs total, drug related and leading to treatment interruption/change
Tolerability (number and proportion of AEs) | 48 weeks
  AEs total, drug related and leading to treatment interruption/change
Bone mineral density | 24 weeks
  change in bone stiffness
Bone mineral density | 48 weeks
  change in bone stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Antiviral Therapy Unit, Ospedali Riuniti, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maggiolo F, Gianotti N, Comi L, Di Filippo E, Fumagalli L, Nozza S, Galli L, Valenti D, Rizzi M, Castagna A. Rilpivirine plus cobicistat-boosted darunavir as alternative to standard three-drug therapy in HIV-infected, virologically suppressed subjects: Final results of the PROBE 2 trial. Antivir Ther. 2021 May;26(3-5):51-57. doi: 10.1177/13596535211042226. Epub 2021 Oct 27. PMID 35485333
- [Derived] Maggiolo F, Gianotti N, Comi L, Di Filippo E, Fumagalli L, Nozza S, Galli L, Valenti D, Rizzi M, Castagna A. Rilpivirine plus cobicistat-boosted darunavir as a two-drug switch regimen in HIV-infected, virologically suppressed subjects on steady standard three-drug therapy: a randomized, controlled, non-inferiority trial (PROBE 2). J Antimicrob Chemother. 2020 May 1;75(5):1332-1337. doi: 10.1093/jac/dkaa018. PMID 32129855